CLINICAL TRIAL: NCT02502721
Title: A Randomized, Open-labeled, Oral Dose, Crossover Design Clinical Trial to Evaluate Pharmacokinetics and Safety Between DWC20151 and DWC20152 in Healthy Male Subjects
Brief Title: A Clinical Trial to Evaluate Pharmacokinetics and Safety Between DWC20151 and DWC20152
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DWJ1373001
Record Dates: First submitted 2015-07-12; First posted 2015-07-20 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): To study effect of DWC20151 on DWC20152 PK
  Interventions: Drug: DWC20151
- Part B (Experimental): To study effect of DWC20152 on DWC20151 PK
  Interventions: Drug: DWC20152

INTERVENTIONS:
Drug: DWC20151
  Arms: Part A
Drug: DWC20152
  Arms: Part B

SUMMARY:
A randomized, open-labeled, oral dose, crossover design clinical trial to evaluate pharmacokinetics and safety between DWC20151 and DWC20152 in healthy male subjects.

DETAILED DESCRIPTION:
This study is to evaluate pharmacokinetics and safety between DWC20151 and DWC20152 in healthy male subjects.

Study design is randomized, open-labeled, oral dose, crossover design. This study will conducted with 2 separated part (Part A, Part B).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects (18~55 years)

Exclusion Criteria:

* Who has allergy to investigational product

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 0~72hr
Area under the plasma concentration versus time curve (AUC) | 0~72h

CONTACTS AND LOCATIONS:
Overall Officials: Jinah Jung, Principal Investigator — Busan paik hospital
Locations (1):
- Busan Paik Hospital, Busan, South Korea